CLINICAL TRIAL: NCT04936087
Title: Wheelchair User's Voice- A Longitudinal Study About the Impact of the WHO-8 Steps for Wheelchair Provision in El Salvador
Brief Title: Effects of the WHO 8-step Wheelchair Service Delivery Process on Wheelchair Users in El Salvador: a Cohort Study
Acronym: WUV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Momentum Wheels for Humanity (Other)
Collaborators: University of Pittsburgh (Other); Universidad de El Salvador (Other); Google LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO18010578; CNEIS/2018/043 (Other: Salvadorian National Committee on Research Ethics for Health)
Record Dates: First submitted 2021-06-02; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Wheelchair Users
Keywords: manual wheelchairs; appropriate service delivery; low- and middle-income countries; global health

STUDY DESIGN:
Intervention Model Description: Longitudinal within-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WHO 8-steps (Other): Single group intervention and described in the Intervention section.
  Interventions: Other: The World Health Organization 8 steps for manual wheelchair service delivery

INTERVENTIONS:
Other: The World Health Organization 8 steps for manual wheelchair service delivery — All study participants were provided with a new wheelchair, a wheelchair cushion, and wheelchair services, delivered by trained wheelchair service providers, according to the WHO 8-step wheelchair service delivery process including assessment, fitting, and a 30-minute individual or group training on 7 wheelchair skills, device care, and pressure injury prevention techniques. Additionally, wheelchair maintenance reminders were sent through a text message service (SMS) to a sub-cohort of participants.
  Wheelchair users were provided with one of three different, International Standards Organization (ISO) tested, wheelchair models according to the users' needs and availability: standard, active, and all-terrain models. All wheelchairs were provided with a basic contour cushion made of polyurethane foam. However, whenever a risk of pressure injury was identified for a study participant, wheelchair providers fabricated a pressure-relief cushion.

SUMMARY:
The objective of this study was to test the hypotheses that wheelchair-related health, wheelchair skills, wheelchair use, poverty probability, and quality of life would improve; and that the number of wheelchair repairs required, adverse events, caregiver burden and the level of assistance provided would decrease after the delivery of manual wheelchairs following the World Health Organization (WHO) 8-step service-delivery process.

This was a longitudinal, within-subject study design including 247 manual wheelchair users in El Salvador. The intervention consisted of the WHO 8-step process as well as maintenance reminders. Outcome assessments on wheelchair-related health, wheelchair skills, wheelchair repairs required, adverse events, caregiver burden and the level of assistance, poverty probability, and quality of life were performed via structured interviews at the initial assessment, at wheelchair delivery, and at 3- and 6-month follow-up. Wheelchair use was measured with dataloggers at assessment, delivery and 3-month follow-up.

DETAILED DESCRIPTION:
Ethics approval was granted from the National Committee on Research Ethics for Health in El Salvador (CNEIS/2018/043) and the Institutional Review Board at the University of Pittsburgh (number PRO18010578). Written informed consent was obtained from all participants before implementing study procedures.

All procedures of the study were conducted at 11 different rehabilitation centers, that served as wheelchair service delivery centers, in El Salvador.

A consecutive sampling method was used to select participants using the waitlists at the 11 rehabilitation centers. The investigators recruited wheelchair users and their caregivers.

Following the initial assessment, all participants were placed on a waiting list until wheelchairs and services were available. All study participants were provided with a new wheelchair (standard, active, or all-terrain model), a wheelchair cushion, and wheelchair services, delivered by trained wheelchair service providers, according to the WHO 8-step wheelchair service delivery process including assessment, fitting, and a 30-minute individual or group training on 7 wheelchair skills, device care, and pressure injury prevention techniques.

In addition, all wheelchairs were provided with a basic contour cushion made of polyurethane foam. However, whenever a risk of pressure injury was identified for a study participant, wheelchair providers fabricated a pressure-relief cushion based on the WHO basic wheelchair service guidelines.

Data were collected between January and November 2019, by a group of eight data collectors from the University of El Salvador.

Study participants were interviewed during the wheelchair assessment (about 2 months before wheelchair delivery), at the wheelchair delivery visit, and at 3- and 6-month follow-up visits after wheelchair delivery. Participants who were not able to attend a follow-up visit were interviewed by phone. Data were collected using the following questionnaires and tools translated into Spanish which included demographic, clinical and wheelchair-related questions, wheelchair skills, maintenance patterns, poverty probability, quality of life, and all their health related questions. Data loggers (DLs) were also used to assess number of days of wheelchair use, daily distance traveled, and speed. Caregivers were interviewed to measure caregiver burden at baseline, at 3-month follow-up, and at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for wheelchair users were being a person with a mobility limitation requiring a wheelchair as a primary means of personal mobility, waiting to receive a new wheelchair from any of the participating wheelchair service delivery centers, 18-years of age or older, had the cognitive and verbal abilities required to respond to the study questions or a proxy who could respond on his or her behalf, and had access to a cellphone.
* Inclusion criteria for caregivers were being a person assisting the wheelchair user with activities of daily living (ADL), 18-years of age or older, being the primary caregiver and willing to participate in the study.

Exclusion Criteria:

* Wheelchair users who required postural support to sit upright were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Massachusetts Institute of Technology (MIT)-Wheelchair-related Health Questionnaire | At month 0 (baseline assessment)
  This questionnaire consists of 25 questions developed to identify the reasons, consequences, and medical attention received for injuries related to the use of the wheelchair such as falls during transfers, falls during maneuvering, injuries to the shoulders, elbows, wrists, hands and back.
Massachusetts Institute of Technology (MIT)-Wheelchair-related Health Questionnaire | At wheelchair delivery (approx. 2 months after baseline assessment)
  This questionnaire consists of 25 questions developed to identify the reasons, consequences, and medical attention received for injuries related to the use of the wheelchair such as falls during transfers, falls during maneuvering, injuries to the shoulders, elbows, wrists, hands and back.
Massachusetts Institute of Technology (MIT)-Wheelchair-related Health Questionnaire | 3 months after wheelchair delivery
  This questionnaire consists of 25 questions developed to identify the reasons, consequences, and medical attention received for injuries related to the use of the wheelchair such as falls during transfers, falls during maneuvering, injuries to the shoulders, elbows, wrists, hands and back.
Massachusetts Institute of Technology (MIT)-Wheelchair-related Health Questionnaire | 6 months after wheelchair delivery
  This questionnaire consists of 25 questions developed to identify the reasons, consequences, and medical attention received for injuries related to the use of the wheelchair such as falls during transfers, falls during maneuvering, injuries to the shoulders, elbows, wrists, hands and back.
Wheelchair Skills Test Questionnaire | At month 0 (baseline assessment)
  The Wheelchair Skills Test Questionnaire, (WST-Q), allows assessing the capacity and frequency with which the wheelchair user performs a series of activities safely in their wheelchair. This instrument consists of 34 questions. Answer to the capacity component can be "no" "yes" "yes, with difficulty" and "not possible with this wheelchair". Possible answers to the frequency component are "always" "sometimes" or "never". Wheelchair Skills Capacity Score is reported in percentage, possible percentage scores range from 0-100%. 0% means the participants do not have the capacity to perform any of the wheelchair skills, and 100% means the participan has the capacity to perform all skills without difficulty.
Wheelchair Skills Test Questionnaire | 3 months after wheelchair delivery
  The Wheelchair Skills Test Questionnaire, (WST-Q), allows assessing the capacity and frequency with which the wheelchair user performs a series of activities safely in their wheelchair. This instrument consists of 34 questions. Answer to the capacity component can be "no" "yes" "yes, with difficulty" and "not possible with this wheelchair". Possible answers to the frequency component are "always" "sometimes" or "never". Wheelchair Skills Capacity Score is reported in percentage, possible percentage scores range from 0-100%. 0% means the participants do not have the capacity to perform any of the wheelchair skills, and 100% means the participan has the capacity to perform all skills without difficulty.
Wheelchair Skills Test Questionnaire | 6 months after wheelchair delivery
  The Wheelchair Skills Test Questionnaire, (WST-Q), allows assessing the capacity and frequency with which the wheelchair user performs a series of activities safely in their wheelchair. This instrument consists of 34 questions. Answer to the capacity component can be "no" "yes" "yes, with difficulty" and "not possible with this wheelchair". Possible answers to the frequency component are "always" "sometimes" or "never". Wheelchair Skills Capacity Score is reported in percentage, possible percentage scores range from 0-100%. 0% means the participants do not have the capacity to perform any of the wheelchair skills, and 100% means the participan has the capacity to perform all skills without difficulty.
Number of days of wheelchair use | At month 0 (baseline assessment)
  Number of days of wheelchair use
Daily distance traveled | At month 0 (baseline assessment)
  Measured in meters per day
Average speed | At month 0 (baseline assessment)
  Measured in meters per second
Number of days of wheelchair use | At wheelchair delivery (approx. 2 months after baseline assessment)
  Number of days of wheelchair use
Daily distance traveled | At wheelchair delivery (approx. 2 months after baseline assessment)
  Measured in meters per day
Average speed | At wheelchair delivery (approx. 2 months after baseline assessment)
  Measured in meters per second
Number of days of wheelchair use | 3 months after wheelchair delivery
  Number of days of wheelchair use
Daily distance traveled | 3 months after wheelchair delivery
  Measured in meters per day
Average speed | 3 months after wheelchair delivery
  Measured in meters per second
Poverty Probability Index for El Salvador | At month 0 (baseline assessment)
  Poverty probability
Poverty Probability Index for El Salvador | 6 months after wheelchair delivery
  Poverty probability
WHO Quality of Life Questionnaire - Brief version | At month 0 (baseline assessment)
  WHO Quality of Life Questionnaire - Brief version (WHOQOL-BREF) was developed to measure the quality of life of people. Its design is suitable to be used in different cultural environments with research objectives, policy making, health practices and auditing. WHOQOL-BREF is the reduced version of WHOQOL-100 and allows a complete evaluation when analyzing four fundamental domains, such as: physical, psychological, social relations and environment. It is designed in such a way that it can be answered by the participant with or without assistance. According to the information provided by the WHO, this tool has been shown to have good discriminating validity, content and reliability.
  The WHOQOL-BREF consists of 26 questions, but a question related to sexual activity was eliminated, because it was considered culturally inappropriate.
  The WHOQOL-BREF domains scores ranges from 4 to 20. A lower a score represents a worse outcome.
WHO Quality of Life Questionnaire - Brief version | 6 months after wheelchair delivery
  WHO Quality of Life Questionnaire - Brief version (WHOQOL-BREF) was developed to measure the quality of life of people. Its design is suitable to be used in different cultural environments with research objectives, policy making, health practices and auditing. WHOQOL-BREF is the reduced version of WHOQOL-100 and allows a complete evaluation when analyzing four fundamental domains, such as: physical, psychological, social relations and environment. It is designed in such a way that it can be answered by the participant with or without assistance. According to the information provided by the WHO, this tool has been shown to have good discriminating validity, content and reliability.
  The WHOQOL-BREF consists of 26 questions, but a question related to sexual activity was eliminated, because it was considered culturally inappropriate.
  The WHOQOL-BREF domains scores ranges from 4 to 20. A lower a score represents a worse outcome.

SECONDARY OUTCOMES:
Wheelchair Maintenance Training Questionnaire | At month 0 (baseline assessment)
  The Wheelchair Maintenance Training Questionnaire (WMT-Q) is dedicated to health professionals and users of manual and power wheelchairs. This questionnaire was designed to obtain information about the frequency to which participants performed certain maintenance activities to their wheelchair. For this study only the version for manual wheelchair users was used. WMT-Q has 20 main questions. Possible answers are: "daily" "weekly" "monthly" "quarterly" "annually" "never".
Wheelchair Maintenance Training Questionnaire | 3 months after wheelchair delivery
  The Wheelchair Maintenance Training Questionnaire (WMT-Q) is dedicated to health professionals and users of manual and power wheelchairs. This questionnaire was designed to obtain information about the frequency to which participants performed certain maintenance activities to their wheelchair. For this study only the version for manual wheelchair users was used. WMT-Q has 20 main questions. Possible answers are: "daily" "weekly" "monthly" "quarterly" "annually" "never".
Wheelchair Maintenance Training Questionnaire | 6 months after wheelchair delivery
  The Wheelchair Maintenance Training Questionnaire (WMT-Q) is dedicated to health professionals and users of manual and power wheelchairs. This questionnaire was designed to obtain information about the frequency to which participants performed certain maintenance activities to their wheelchair. For this study only the version for manual wheelchair users was used. WMT-Q has 20 main questions. Possible answers are: "daily" "weekly" "monthly" "quarterly" "annually" "never".
Zarit Burden Interview - short version | At month 0 (baseline assessment)
  The Zarit Caregiver Burden Questionnaire - short version, or better known as ZBI-12 (Zarit Burden Interview), consists of 12 questions that evaluate the burden of caregivers of people with senile dementia and people with disabilities. The ZBI assesses the caregiver's burden taking into account aspects of the caregiver's life such as family, free time and social activities. This questionnaire can be self-administered, has high content validity, high internal consistency, and great confidence of repetition. The ZBI is available in Spanish, so it can was used in El Salvador as an instrument to measure caregiver burden. ZBI Score range: 0 to 48. The higher the score, the greater the burden of care.
Zarit Burden Interview - short version | 3 months after wheelchair delivery
  The Zarit Caregiver Burden Questionnaire - short version, or better known as ZBI-12 (Zarit Burden Interview), consists of 12 questions that evaluate the burden of caregivers of people with senile dementia and people with disabilities. The ZBI assesses the caregiver's burden taking into account aspects of the caregiver's life such as family, free time and social activities. This questionnaire can be self-administered, has high content validity, high internal consistency, and great confidence of repetition. The ZBI is available in Spanish, so it can was used in El Salvador as an instrument to measure caregiver burden. ZBI Score range: 0 to 48. The higher the score, the greater the burden of care.
Zarit Burden Interview - short version | 6 months after wheelchair delivery
  The Zarit Caregiver Burden Questionnaire - short version, or better known as ZBI-12 (Zarit Burden Interview), consists of 12 questions that evaluate the burden of caregivers of people with senile dementia and people with disabilities. The ZBI assesses the caregiver's burden taking into account aspects of the caregiver's life such as family, free time and social activities. This questionnaire can be self-administered, has high content validity, high internal consistency, and great confidence of repetition. The ZBI is available in Spanish, so it can was used in El Salvador as an instrument to measure caregiver burden. ZBI Score range: 0 to 48. The higher the score, the greater the burden of care.
Checklist of Activities of Daily Living | At month 0 (baseline assessment)
  The checklist of Activities of Daily Living is a questionnaire designed to collect information about the level of assistance provided to wheelchair users by caregivers in 17 activities of daily living. Possible responses are "Requires no assistance" "Some assistance needed" "Complete assistance needed" and "Not applicable". Responses are reported in number of activities under each level of assistance.
Checklist of Activities of Daily Living | 3 months after wheelchair delivery
  The checklist of Activities of Daily Living is a questionnaire designed to collect information about the level of assistance provided to wheelchair users by caregivers in 17 activities of daily living. Possible responses are "Requires no assistance" "Some assistance needed" "Complete assistance needed" and "Not applicable". Responses are reported in number of activities under each level of assistance.
Checklist of Activities of Daily Living | 6 months after wheelchair delivery
  The checklist of Activities of Daily Living is a questionnaire designed to collect information about the level of assistance provided to wheelchair users by caregivers in 17 activities of daily living. Possible responses are "Requires no assistance" "Some assistance needed" "Complete assistance needed" and "Not applicable". Responses are reported in number of activities under each level of assistance.
Breakdowns and Adverse Consequences Questionnaire | At month 0 (baseline assessment)
  The Breakdowns and Adverse Consequences Questionnaire (BAC-Q) allows to collect information about the failures that occurred in the wheelchairs. BAC-Q allows knowing the failures in the tires, front wheels, the wheelchair frame, elements of postural support, seat, backrest, cushion, and it gives the opportunity to indicate another type of failure if necessary. By means of this questionnaire it is possible to know the person who carried out the repair and the consequences in the users due to wheelchair breakdowns. For example, being stranded at home or away from home, injuries due to failure, lack of school attendance, work, medical appointments, or other.
Breakdowns and Adverse Consequences Questionnaire | At wheelchair delivery (approx. 2 months after baseline assessment)
  The Breakdowns and Adverse Consequences Questionnaire (BAC-Q) allows to collect information about the failures that occurred in the wheelchairs. BAC-Q allows knowing the failures in the tires, front wheels, the wheelchair frame, elements of postural support, seat, backrest, cushion, and it gives the opportunity to indicate another type of failure if necessary. By means of this questionnaire it is possible to know the person who carried out the repair and the consequences in the users due to wheelchair breakdowns. For example, being stranded at home or away from home, injuries due to failure, lack of school attendance, work, medical appointments, or other.
Breakdowns and Adverse Consequences Questionnaire | 3 months after wheelchair delivery
  The Breakdowns and Adverse Consequences Questionnaire (BAC-Q) allows to collect information about the failures that occurred in the wheelchairs. BAC-Q allows knowing the failures in the tires, front wheels, the wheelchair frame, elements of postural support, seat, backrest, cushion, and it gives the opportunity to indicate another type of failure if necessary. By means of this questionnaire it is possible to know the person who carried out the repair and the consequences in the users due to wheelchair breakdowns. For example, being stranded at home or away from home, injuries due to failure, lack of school attendance, work, medical appointments, or other.
Breakdowns and Adverse Consequences Questionnaire | 6 months after wheelchair delivery
  The Breakdowns and Adverse Consequences Questionnaire (BAC-Q) allows to collect information about the failures that occurred in the wheelchairs. BAC-Q allows knowing the failures in the tires, front wheels, the wheelchair frame, elements of postural support, seat, backrest, cushion, and it gives the opportunity to indicate another type of failure if necessary. By means of this questionnaire it is possible to know the person who carried out the repair and the consequences in the users due to wheelchair breakdowns. For example, being stranded at home or away from home, injuries due to failure, lack of school attendance, work, medical appointments, or other.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Pearlman, Principal Investigator — University of Pittsburgh
Locations (13):
- El Salvador (13):
  - Foundation Pro Rehabilitation Teleton- FUNTER Merliot, Antiguo Cuscatlán
  - Medical Unit Ilopango -ISSS, Ilopango
  - Polyclinic Hospital Planes de Renderos -ISSS, Planes de Renderos
  - Regional Hospital San Miguel -ISSS, San Miguel
  - Medical Unit 15 de Septiembre -ISSS, San Salvador
  - Physical Medicine and Rehabilitation Unit- ISSS, San Salvador
  - Foundation Pro Rehabilitation Teleton- FUNTER San Vicente, San Vicente
  - Santa Ana's Hospital -ISSS, Santa Ana
  - El Salvador's UCP Wheels for Humanity, Santa Tecla
  - Foundation Pro Rehabilitation Teleton- FUNTER Sonsonate, Sonsonate
  - Sonsonate's Regional Hospital -ISSS, Sonsonate
  - Usulutan's Hospital -ISSS, Usulután
  - Polyclinic Hospital Zacamil -ISSS, Zacamil

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IDP), all IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Starting after publication
Access Criteria: All data files will be available from the Inter-university Consortium for Political and Social Research (ICPSR) database. Students, researchers, instructors, staff, and everyone else affiliated with a member institution receives full access to all of ICPSR's data.
URL: https://www.icpsr.umich.edu/web/pages/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04936087/Prot_SAP_000.pdf